CLINICAL TRIAL: NCT01090271
Title: Eccentric Training for Shoulder Abductors Improves Pain, Function and Isokinetic Performance Steadiness in Subjects With Shoulder Impingement Syndrome
Brief Title: Effects of Eccentric Training for Shoulder Abductors in Subjects With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenaçao de Aperfeiçoamento de Pessoal de Nível Superior (Unknown)
Responsible Party: Tânia de Fátima Salvini, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UFSCar-214/2007
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2007-09

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Subacromial impingement syndrome; Muscle Strength; Resistance Training
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eccentric training (Experimental)
  Interventions: Device: Isokinetic eccentric training

INTERVENTIONS:
Device: Isokinetic eccentric training — The eccentric training for the shoulder abductors was performed for 6 consecutive weeks, twice a week, on alternate days.

SUMMARY:
The aim of the study was to evaluate the effect of eccentric strength training for shoulder abductors on force steadiness in subjects with subacromial impingement syndrome (SIS).

DETAILED DESCRIPTION:
Although it is known that shoulder abduction in subjects with subacromial impingement syndrome (SIS) presents alterations in several parameters, as for example, in scapular and glenohumeral kinematics, the strengthening of the shoulder abductors as an intervention strategy is controversial in literature.

Strength training has been shown to be effective in reducing the fluctuations in force and had a positive effect on isometric steadiness in old adults and in healthy young subjects during bed rest. However, there are no studies that evaluated the effects of strength training on the force steadiness in subjects with SIS.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with Subacromial impingement syndrome by a physical therapist (the diagnosis was confirmed by an orthopaedic physician).

Exclusion Criteria:

* pregnancy
* torn rotator cuff or long head biceps tendons
* ligamentous laxity based on positive Sulcus test or a positive apprehension test
* previous shoulder or neck surgery
* hooked acromion
* systemic illnesses
* corticosteroid injection 3 months prior to evaluation
* physical therapy 6 months prior to evaluation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Isokinetic evaluation | 2 months

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Tânia TS Salvini, PhD, Principal Investigator — Universidade Federal de Sao Carlos (Sao Paulo - Brazil)
Locations (1):
- Universidade Federal de Sao Carlos, São Carlos, São Paulo, Brazil